CLINICAL TRIAL: NCT06333405
Title: Evaluation of the Safety of Fecal Microbiota Transplantation (FMT) as a Prophylaxis of Necrotizing Enterocolitis (NEC) in a Group of Newborns at Increased Risk for the Disease
Brief Title: Fecal Microbiota Transplantation (FMT) as a Prophylaxis of Necrotizing Enterocolitis (NEC) - Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FMTNEC/01/2024
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Necrotizing Enterocolitis
Keywords: Enterocolitis, Necrotizing; Fecal Microbiota Transplantation; Necrotizing Enterocolitis prophylaxis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Enterocolitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: single group, open label, observational study with intervention (FMT)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Fecal Microbiota Transplantation (Experimental)
  Interventions: Drug: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Procedure: Fecal Microbiota Transplantation
  Fecal Microbiota as a suspension obtained from healthy unrelated donor (woman in 3rd trimester of pregnancy) introduced two times per treatment:
  * as a deep rectal infusion, via Foley's catheter inserted under ultrasound control, twice 6 hours apart, between 3 and 6 days after birth and/or up to 14 days
  * Other Names: MBiotix HBI

SUMMARY:
The aim of the study is to assess the safety of fecal microbiota transplantation (FMT) as a preventive method for the development of Necrotizing enterocolitis (NEC) in a group of premature infants.

This is the first stage of a clinical trial testing the effectiveness of FMT in NEC, the aim of which is to examine the safety profile and analyze all side effects.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is an inflammatory disease with an incidence of about 1 in 1,000 live births, much higher in premature and low birth weight newborns. Mortality in this disease reaches about 15-30% and has remained stable for many years. Intestinal dysbiosis is an important element of the pathogenesis of this disease and for this reason, experimental models have been used to administer fecal microbiota transplantation (FMT) for prophylaxis and treatment of NEC with very satisfactory results. The aim of the study is to investigate the safety of FMT in the prophylaxis of NEC in premature neonates.

FMT preparation will be prepared specifically for this study by the Human Biome Institute (HBI), with which a scientific collaboration has been established for this experiment. The donors of the material from which the FMT will be prepared will be women in the third trimester of pregnancy who will consent to the collection the material from them, and who will pass a detailed health questionnaire and medical and additional examinations in accordance with the donor qualification protocol according to international recommendations in the method and the procedure developed by the HBI (Human Biome Institute).

During this interventional, prospective, single arm, open-label, observational study, the investigators will collect the information about the safety of FMT in the prophylaxis of NEC.

The project protocol is based on the intervention (fecal microbiota transplantation; FMT) as a deep rectal infusion, via Foley's catheter inserted under ultrasound control. The procedure will be conducted twice, 6 hours apart, between 3 and 6 days after birth and/or up to 14 days, to participants who have transient contraindications to FMT or to participants who will be referred for treatment at our facility from an outpatient facility.

After the procedure, the participants will be closely monitored for adverse reactions up to the discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants hospitalized in the intensive care unit and neonatal pathology unit during the study period

  1. 1. Born naturally or by cesarean section between:

     1. 24 0/7 and 36 6/7 weeks of gestation
  2. Age >48 hours, a minimum of 24 hours after completion of antibiotic therapy and up to day 14 for newborns <35 weeks of gestation and up to day 6 for newborns >35 weeks of gestation
  3. Newborns born in and out of hospital
  4. Parental consent to participate in the study

Exclusion Criteria:

1. Occurrence of congenital defects of the gastrointestinal tract preventing proper intestinal passage (esophageal atresia, duodenal atresia, rectal atresia, tracheo-esophageal fistulas) and occurrence of genetic diseases diagnosed prenatally or at birth (trisomies, other genetic syndromes).
2. Gastrointestinal perforation
3. Food allergy with anaphylactic shock
4. Participation in another clinical trial that may affect the final outcome of the planned intervention

Temporary exclusion criteria

If at least 1 of the following occurs before FMT and up to 14 days of age:

1. Intolerance to oral feeding, based on the assessment of the qualifying physician on the day of FMT:

   * painful bloating in the abdomen and/or visible bowel loops, blood in the stools,
   * delayed gastric emptying: two consecutive episodes exceeding >50% of the volume of the previous serving, 2 or more consecutive episodes of retention / vomiting / regurgitation of biliary contents / duodenal contents/ blood - episodes not related to anxiety, delayed bowel movements, possibility of swallowing blood during childbirth or from damaged nipples, abnormality of the positioning of gastric tube, bleeding from the nose
2. Suspected NEC:

   * clinical signs typical for NEC - Bell criteria, redness/bruising of the anterior abdominal wall, palpable abdominal resistance, hypotension; laboratory signs: hyponatraemia, metabolic acidosis, thrombocytopenia, increased inflammation parameters)
3. Antibiotic therapy during planned FMT treatment
4. Clinical signs of infection or significantly elevated inflammatory parameters - If at least one of the following clinical signs and/or more than 1 laboratory sign occurs:

   • Clinical signs of infection: Hemodynamic instability (hypotension, tachycardia, peripheral circulatory disturbances (by age standards), thermoregulatory disturbances, fever>38 deg C, hypothermia <36 deg C) Apathy, lethargy, convulsions Apneas, deterioration of respiratory capacity

   • Labolatory signs of infection:

   Elevated inflammatory parameters:
   * leukocytosis <5 i >30x109/L up to 48 hours of life (HoL) and <5 i >20x109/L >48 hours of life, the band neutrophil : total neutrophil (I:T) ratio of >0.2 for >34 weeks of gestation and >0,16 for <34 weeks of gestation
   * CRP >0.05mg/l (at the norm up to <0.05-1mg/l),
   * PCT (>72 HoL) > 0,5-1ng/ml (at the norm up to > 0,5-1ng/ml); Platelet count < 50K, coagulopathy positive cultures of normally sterile body fluids

     * Radiological evidence of infection, including systemic e. g. gallbladder bed swelling, unexplained sudden echocardiographic pulmonary hypertension

Ages: 24 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions monitoring | Up to the discharge from the hospital (approximately from 2 weeks to 3 months)
  The safety of the procedure will be assessed on the basis of:
  1. number of episodes of oral feeding intolerance, diarrhoea, blood/mucus/pus in stools
  2. appearance of symptoms of infection or significant change in vital parameters (heart rate ECG and oxygen saturation - continuous measurement, blood pressure 4x/day, temperature, possibly HERO)
  3. number of developed NEC
  4. assessment of blood flow in the upper mesenteric artery by ultrasound
  5. observation of other symptoms - convulsions, unbridled crying, anxiety
  6. the number of positive blood cultures, the percentage of antibiotic therapy
  7. number of serious side effects - death, serious threat to health and/or life and/or deterioration of health
  8. Length of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Pediatric Surgery Clinic, Warsaw, Mazovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prado C, Michels M, Avila P, Burger H, Milioli MVM, Dal-Pizzol F. The protective effects of fecal microbiota transplantation in an experimental model of necrotizing enterocolitis. J Pediatr Surg. 2019 Aug;54(8):1578-1583. doi: 10.1016/j.jpedsurg.2018.10.045. Epub 2018 Oct 22. PMID 30414693
- [Background] Liu J, Miyake H, Zhu H, Li B, Alganabi M, Lee C, Pierro A. Fecal microbiota transplantation by enema reduces intestinal injury in experimental necrotizing enterocolitis. J Pediatr Surg. 2020 Jun;55(6):1094-1098. doi: 10.1016/j.jpedsurg.2020.02.035. Epub 2020 Feb 26. PMID 32234317
- [Background] Li X, Li X, Shang Q, Gao Z, Hao F, Guo H, Guo C. Fecal microbiota transplantation (FMT) could reverse the severity of experimental necrotizing enterocolitis (NEC) via oxidative stress modulation. Free Radic Biol Med. 2017 Jul;108:32-43. doi: 10.1016/j.freeradbiomed.2017.03.011. Epub 2017 Mar 16. PMID 28323128
- [Background] Hui Y, Vestergaard G, Deng L, Kot WP, Thymann T, Brunse A, Nielsen DS. Donor-dependent fecal microbiota transplantation efficacy against necrotizing enterocolitis in preterm pigs. NPJ Biofilms Microbiomes. 2022 Jun 9;8(1):48. doi: 10.1038/s41522-022-00310-2. PMID 35680942
- [Background] Korpela K, Helve O, Kolho KL, Saisto T, Skogberg K, Dikareva E, Stefanovic V, Salonen A, Andersson S, de Vos WM. Maternal Fecal Microbiota Transplantation in Cesarean-Born Infants Rapidly Restores Normal Gut Microbial Development: A Proof-of-Concept Study. Cell. 2020 Oct 15;183(2):324-334.e5. doi: 10.1016/j.cell.2020.08.047. Epub 2020 Oct 1. PMID 33007265
- [Background] Ma X, Xu T, Qian M, Zhang Y, Yang Z, Han X. Faecal microbiota transplantation alleviates early-life antibiotic-induced gut microbiota dysbiosis and mucosa injuries in a neonatal piglet model. Microbiol Res. 2022 Feb;255:126942. doi: 10.1016/j.micres.2021.126942. Epub 2021 Dec 10. PMID 34915267